CLINICAL TRIAL: NCT05689359
Title: Phase 2, Single Center, Single Arm Study to Evaluate the Decrease in CIPN With the Addition of Hydroxychloroquine to Chemotherapy in Patients With Early Stage (1-3) Breast Cancer and Gynecological Cancers Treated With Curative Intent
Brief Title: Evaluation of Hydroxychloroquine to Prevent CIPN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Per Principal Investigator, it is not feasible to move forward with this trial.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001721
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Gynecologic Cancer; Early-stage Breast Cancer; Peripheral Neuropathy; Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy Induced Peripheral Neuropathy; Hydroxycloroquine; Diffusion Tensor Imaging; Breast Cancer; Gynecologic Cancer; Paclitaxel; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Addition of Hydroxychloroquine to paclitaxel (Experimental): Hydroxychloroquine will be added to chemotherapy in patients with early stage (1-3) breast cancer and gynecological cancers.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine will be administered at 600 mg po BID for 3 days prior to starting chemotherapy, continued during the course of chemotherapy, and for 7 days after chemotherapy.

SUMMARY:
The study is being done to research if hydroxychloroquine can prevent chemotherapy induced peripheral neuropathy. Certain chemotherapy drugs, like paclitaxel, are known to cause neuropathy which can impact quality of life. Currently, there are no options for preventing peripheral neuropathy. In addition, there are no useful methods to assess peripheral nerve damage. This study will also explore using a study MRI of patients' feet prior to starting chemotherapy and after they have completed chemotherapy to see if there is any difference in their nerve structure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 1-3 breast cancer or gynecological cancer treated with curative intent
* Age ≥ 21 years old
* No prior neurotoxic chemotherapies
* No other neurotoxic chemotherapies planned during paclitaxel treatment (i.e, platinum)
* Need to be treated with paclitaxel weekly x 12 doses as determined by their treating physician
* Be able to undergo MR Imaging
* Be willing to comply with scheduled visits, treatment plan, and MR imaging
* Adequate organ function as defined as:

Hematologic:

Absolute neutrophil count (ANC) ≥ 1500/mm3 Platelet count ≥ 100,000/mm3 Hemoglobin ≥ 9 g/dL

Hepatic:

Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN

Renal:

Estimated creatinine clearance (CrCl)≥ 50 mL/min by Cockcroft-Gault formula

Exclusion Criteria:

* Stage IV cancer
* CTCAE neurological function > grade 1 at baseline
* Mental limitation that precludes understanding of or completion of questionnaires
* History of diabetes or other neurological disorders
* Preexisting peripheral neuropathy
* Prior exposure to neurotoxic chemotherapy
* Currently taking medication to treat or prevent neuropathy
* Have non-MRI compatible metallic objects on/in body
* Have metallic hardware in the lower extremity which is MR compatible however would create too much artifact for MR examination
* Pregnant or lactating patients. Women of childbearing potential and sexually active men must use an effective contraception method during rreatment and for three months after completing treatment. Patients of childbearing potential must have a negative serum or urine B-hCG pregnancy test at screening.
* History or current evidence of central serous retinopathy (CSR) or retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity) or macular degeneration.
* QTc prolongation defined as a QTcF > 500 ms
* Known glucose-6-phosphate dehydrogenase (G-6-PD) deficiency.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Symptomatic CIPN | Throughout study completion, an average of 6 months
  The primary endpoint is symptomatic CIPN defined as increase in in FACT-GOG/Ntx-12 questionnaire score of greater than or equal to 3 points post-chemotherapy with hydroxychloroquine in combination with paclitaxel chemotherapy in patients with early-stage breast cancer or gynecologic malignancies.

SECONDARY OUTCOMES:
Predicting Symptomatic CIPN: FA and ADC values derived from DTI | Baseline
  Baseline fractional anisotrophy (FA) and apparent diffusion coefficient (ADC) values derived from DTI will be used to predict symptomatic CIPN prior to starting and end of chemotherapy.
Predicting Symptomatic CIPN: change in FA and ADC | Baseline and 12 weeks
  Change in mean FA and ADC prior to starting and end of chemotherapy will be calculated. The mean of the change in FA and ADC values with 95% confidence intervals will be estimated (post- minus pre- chemotherapy). The baseline values and the change of FA and ADC will be used to predict the development of symptomatic CIPN using logistic regression.
Predicting Symptomatic CIPN: baseline NF-L levels | Baseline
  Baseline level of neurofilament light chain (NF-L) will be used to predict symptomatic CIPN. The baseline values will be used to predict development of symptomatic CIPN using logistic regression.
Predicting Symptomatic CIPN: Changes in NF-L levels | Baseline and 12 weeks
  Changes in NF-L levels with chemotherapy used to predict development of symptomatic CIPN. NF-L measures will be summarized across time and analyzed using linear mixed effects model.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Segar, MD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No